CLINICAL TRIAL: NCT00004333
Title: Phase II Study of the Enzyme Inhibitor NTBC for Tyrosinemia Type I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Michigan (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11892; UMMC-1319
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-07

CONDITIONS: Tyrosinemia, Type I
Keywords: inborn errors of metabolism; rare disease; tyrosinemia I
MeSH Terms: conditions — Tyrosinemias; Metabolism, Inborn Errors; Rare Diseases

INTERVENTIONS:
Drug: NTBC

SUMMARY:
OBJECTIVES:

Assess whether 2-(2-nitro-4-trifluoromethylbenzoyl)-1,3-cyclohexanedione (NTBC) at 0.6 mg/kg per day prevents liver failure in at least 1 patient with tyrosinemia type I.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Only 2 patients with tyrosinemia type I are known to this research team; others will be treated if found and if clinical conditions permit.

The enzyme inhibitor 2-(2-nitro-4-trifluoromethylbenzoyl)-1,3-cyclohexanedione (NTBC) is administered orally, in 2 divided doses daily with meals.

Patients will be followed closely for side effects attributable to NTBC.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Tyrosinemia type I No cirrhosis No hepatocellular carcinoma

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-11

CONTACTS AND LOCATIONS:
Overall Officials: Jess G. Thoene, Study Chair — University of Michigan